CLINICAL TRIAL: NCT05666154
Title: Targeted Elimination Diet in FD Patients Following Identification of Trigger Nutrients Using Confocal Laser Endomicroscopy
Brief Title: Confocal Laser Endomicroscopy Based Diet in Functional Dyspepsia
Acronym: CLEFD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S65735
Record Dates: First submitted 2021-12-09; First posted 2022-12-27 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Functional Dyspepsia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Real diet (Active Comparator): Diet excluding the trigger nutrient identified by an acute mucosal reaction in CLE
  Interventions: Other: Real diet
- Sham diet (Sham Comparator): Diet excluding a sham nutrient without acute mucosal reaction in CLE
  Interventions: Other: Sham diet
- Wheat exclusion diet (Active Comparator): In patients without identified trigger nutrient (i.e. no acute mucosal reaction to any nutrient), wheat will be excluded as an empirical diet in crossover fashion with soy.
  Interventions: Other: Wheat exclusion diet
- Soy exclusion diet (Active Comparator): In patients without identified trigger nutrient (i.e. no acute mucosal reaction to any nutrient), wheat will be excluded as an empirical diet in crossover fashion with soy.
  Interventions: Other: Soy exclusion diet

INTERVENTIONS:
Other: Real diet — Diet excluding either trigger nutrient in a blinded crossover fashion (CLE positive individuals with identified trigger)
  Arms: Real diet
Other: Sham diet — Diet excluding either sham nutrient in a blinded crossover fashion (CLE positive individuals with identified trigger) or wheat and soy in a blinded crossover fashion (CLE negative individuals without identified trigger)
  Arms: Sham diet
Other: Wheat exclusion diet — Diet excluding wheat in a blinded crossover fashion (CLE negative individuals without identified trigger)
  Arms: Wheat exclusion diet
Other: Soy exclusion diet — Diet excluding soy in a blinded crossover fashion (CLE negative individuals without identified trigger)
  Arms: Soy exclusion diet

SUMMARY:
After a thorough baseline evaluation, functional dyspepsia (FD) patients will be exposed to nutrients while undergoing confocal laser endomicroscopy (CLE). Patients presenting an acute mucosal reaction upon nutrient exposure will be instructed to exclude their respective trigger nutrient or a nutrient without mucosal reaction (=sham diet) from their diet for 4 weeks in a randomized, blinded crossover fashion.

The aim of the trial is to assess the symptomatic response to the targeted diet and further elucidate mechanisms underlying the acute mucosal reactions observed in CLE upon nutrient exposure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 y/o (70 years included)
* Male or female subjects
* FD (PDS, EPS or overlap) according to Rome IV criteria
* Provide written informed consent to participate in the study
* Women of child-bearing potential agree to apply a highly effective method of birth control during the entire duration of the trial. Highly effective birth control is defined as those which result in a low failure rate (i.e., less than 1% per year) when used constantly and correctly such as implants, injectables, combined oral contraceptive method, or some intrauterine devices (IUDs), sexual abstinence, or vasectomized partner. Women of non-childbearing potential may be included if surgically sterile (tubal ligation or hysterectomy) or postmenopausal with at least 2 year without spontaneous menses.
* Subjects who are capable to understand the study and the questionnaires, and to comply with the study requirements.

Exclusion Criteria:

* Pregnant or breastfeeding women
* History of major surgery of the gastrointestinal tract (cholecystectomy and uncomplicated appendectomy are allowed)
* Symptoms predominantly associated with irritable bowel syndrome or gastro-esophageal reflux disease
* IgE-mediated food allergies identified by immunocaps blood tests
* Known underlying organic gastrointestinal disease
* Current use of NSAIDs, proton-pump inhibitors, systemic histamine-receptor antagonists, mast cell stabilizers, corticosteroids, opioids (need to be stopped at least 2 weeks). Use of antibiotics in the past 6 weeks.
* Allergy to Fluorescein or Propofol
* Known celiac disease
* Following a diet, interfering with the study diet in opinion to the investigators

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2021-12-05 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Responder rates in targeted diet vs sham diet | After 4 weeks of dietary intervention
  Response defined by an improvement of minimum 0.5 points on the LPDS scale

SECONDARY OUTCOMES:
Baseline duodenal transepithelial electrical resistance between groups | At baseline
  Differences in baseline permeability measures (TEER and flux, measured with ussing chambers on duodenal biopsies) between CLE positive and negative patients and healthy volunteers using Ussing chambers
Baseline duodenal flux of horse-radish peroxidase between groups | At baseline
  Differences in baseline permeability measures (flux, measured with ussing chambers on duodenal biopsies) between CLE positive and negative patients and healthy volunteers using Ussing chambers
Evolution of duodenal flux of horse-radish peroxidase between dietary interventions | Baseline and after 4 weeks of diet
  Differences in permeability measures (HRP flux, measured with ussing chambers on duodenal biopsies) between dietary interventions (i.e. verum, sham, wheat and soy) during the dietary interventions using urinary Lactulose/Mannitol/Sucralose ratio
Evolution of duodenal transepithelial electrical resistance between dietary interventions | Baseline and after 4 weeks of diet
  Differences in permeability measures (TEER, measured with ussing chambers on duodenal biopsies) between dietary interventions (i.e. verum, sham, wheat and soy) during the dietary interventions using urinary Lactulose/Mannitol/Sucralose ratio
Baseline mucosal immune cell composition between groups | Baseline
  Differences in baseline mucosal mast-cell and eosinophil counts between CLE positive and negative patients

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided